CLINICAL TRIAL: NCT02867891
Title: Multicenter, Observational Trial to Determine the Response Rate of Sorafenib and Donor Lymphocyte Infusions (DLI) Versus Best Available Treatment (BAT) in FLT3-ITD-mutant AML Relapse After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Sorafenib In Relapse of FMS-like Tyrosine Kinase 3 (FLT3)-Internal Tandem Duplication (ITD) AML Trial
Acronym: SIRA
Status: Completed | Type: Observational
Sponsor: Robert Zeiser (Other)
Responsible Party: Sponsor-Investigator, Robert Zeiser, Head of Tumor Imunnology and Immun regulation, University of Freiburg
Organization: University of Freiburg (Other)
Other Study IDs: SIRA
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: FLT3-ITD; AML; allo-HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum cytokine levels (IL-15, IFN-gamma, IL-6)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Chemotherapy alone: The specific interventions to the subjects of the study are assigned by the individual transplant center
- Chemotherapy/DLI: The specific interventions to the subjects of the study are assigned by the individual transplant center
- Sorafenib alone: The specific interventions to the subjects of the study are assigned by the individual transplant center
- Sorafenib/DLI: The specific interventions to the subjects of the study are assigned by the individual transplant center

SUMMARY:
In this trial the investigators will evaluate the outcomes of 4 pre-defined groups of individuals according to the therapeutic intervention. The investigators will determine the outcome of each group by monitoring the survival and the response rates of patients with FLT3-ITD AML relapse after allo-HSCT.

DETAILED DESCRIPTION:
The preliminary data of the investigators demonstrate potent activity of Sorafenib combined with Donor lymphocyte infusions (DLI) in relapse of FLT3-ITD+ Acute myeloid leukemia (AML) after allogeneic hematopoietic cell transplantation (allo-HSCT). The investigators therefore launched an observational multicenter trial. The outcomes are assessed in 4 pre-defined groups of individuals according to the therapeutic intervention (chemotherapy-alone-group, chemotherapy/DLI group, sorafenib alone group and sorafenib/DLI group). The specific interventions to the subjects of the study are assigned by the individual transplant center. The investigators will determine the outcome of each group by monitoring the survival and the response rates (complete remission, disease burden reduction, no response) of patients with FLT3-ITD AML relapse after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Histology/PCR proven relapse of FLT3-ITD+ AML after allo-HSCT
* Age ≥18 years
* Treatment with either chemotherapy-alone, chemotherapy/DLI, sorafenib alone or sorafenib/DLI
* Written informed consent
* Ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* Age < 18 years
* Lack of informed consent
* Patients that cannot be classified in one of the 4 groups: chemotherapy-alone-group, chemotherapy/DLI group, sorafenib alone group and sorafenib/DLI group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapse of FLT3-ITD AML after allogeneic hematopoietic stem cell transplantation
Sampling Method: Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2001-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 10 years
  The primary endpoint is response to treatment, defined as the number of participants that archive a complete remission.

SECONDARY OUTCOMES:
Overall survival (OS) of the participants | 10 years
Serum cytokine levels (Interleukin (IL)-15, Interferon-gamma, IL-6) of the participants. | 10 years
Number of participants with acute graft-versus-host disease (GvHD). | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — Medical Center University of Freiburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metzelder SK, Schroeder T, Finck A, Scholl S, Fey M, Gotze K, Linn YC, Kroger M, Reiter A, Salih HR, Heinicke T, Stuhlmann R, Muller L, Giagounidis A, Meyer RG, Brugger W, Vohringer M, Dreger P, Mori M, Basara N, Schafer-Eckart K, Schultheis B, Baldus C, Neubauer A, Burchert A. High activity of sorafenib in FLT3-ITD-positive acute myeloid leukemia synergizes with allo-immune effects to induce sustained responses. Leukemia. 2012 Nov;26(11):2353-9. doi: 10.1038/leu.2012.105. Epub 2012 Apr 16. PMID 22504140
- [Background] De Freitas T, Marktel S, Piemontese S, Carrabba MG, Tresoldi C, Messina C, Lupo Stanghellini MT, Assanelli A, Corti C, Bernardi M, Peccatori J, Vago L, Ciceri F. High rate of hematological responses to sorafenib in FLT3-ITD acute myeloid leukemia relapsed after allogeneic hematopoietic stem cell transplantation. Eur J Haematol. 2016 Jun;96(6):629-36. doi: 10.1111/ejh.12647. Epub 2015 Sep 21. PMID 26260140